CLINICAL TRIAL: NCT01005849
Title: A Parallel, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Probiotic Formula in the Prevention of Traveler's Diarrhea
Brief Title: Probiotics and the Prevention of Traveler's Diarrhea
Acronym: TD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: because of low rate recruitment and the inability to reach the target expected
Sponsor: Lallemand SAS (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Dr. Henri Durand, Scientific Director, Lallemand SAS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #09-prot-2-lal-01
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-03

CONDITIONS: Travelers' Diarrhea
Keywords: Probiotics; Traveler's diarrhea; Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protecflor (Experimental)
  Interventions: Dietary Supplement: Protecflor
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protecflor — 1 Capsule to be taken once a day during the entire study period
  Arms: Protecflor
Dietary Supplement: Placebo — 1 Capsule to be taken once a day during the entire study period
  Arms: Placebo

SUMMARY:
The present study is designed to evaluate the effect of a mixture of probiotics on the prevention of traveler's diarrhea (TD) in subjects who travel to a country with a high risk for developing TD. Subjects will be asked to take one capsule containing a mixture of probiotics or a placebo capsule a day, within the week before departure, during the travel and up to 3 days after return. They will note the following outcomes in a diary: occurence of diarrhea, number and consistency of stools, duration of the diarrhea, presence of diarrhea-related symptoms and need for rescue medication.

The present study will examine if the use of the probiotics capsule reduces the occurence of traveler's diarrhea as compared to the placebo capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 or over. Upper age limit set by subject's ability to participate in the study;
2. Subject must give written informed consent;
3. Plan to travel to a geographic area with high risk of TD with a travel duration between 12 and 14 days;
4. Subjects must be willing to refrain from using anti-diarrheal medications or antibiotics during the study period, unless they become clinically indicated in which case a rescue regimen can be administered;
5. Subjects willing to refrain from eating yoghurt and taking other probiotics during the study;
6. Female subjects of child-bearing potential must agree to use adequate birth control during the study period. This will be defined as hormonal contraception or a double barrier-method.

Exclusion Criteria:

1. Subjects who have been previously treated with PROTECFLOR® or who have participated in previous Lallemand-sponsored studies;
2. Subjects who have been born in a developing country.
3. Subjects with a history of substance or alcohol abuse or any other psychological condition that may, in the investigator's opinion, adversely affect their co-operation with the study;
4. Subjects who receive a cholera vaccine
5. Subjects with chronic diarrhea;
6. Subjects with chronic disease such as irritable bowel syndrome (IBS) or inflammatory bowel disease (IBD) or ulcerative colitis (UC) ;
7. Subjects with gastrointestinal (GI) surgery during the last 3 months;
8. Subjects who took systemic antibiotic 15 days or less prior to the study;
9. Subjects with immunodeficiency's or immune suppression;
10. Subjects being treated for cancer with radiotherapy and/or chemotherapy;
11. Subjects with organ transplants;
12. Subjects treated with immunosuppressant drugs;
13. Subjects receiving another probiotic preparations or having received probiotic preparations within the last 15 days;
14. Subjects with tube feeding, ileostomy and colostomy;
15. Subjects diagnosed Clostridium difficile colitis within the last 3 months;
16. Women who are pregnant, or who will not consent to using adequate birth control during the study period;
17. Women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Occurence of traveler's diarrhea | 3 weeks

SECONDARY OUTCOMES:
Number and consistency of stools (normal, soft or unformed) | 3 weeks
Duration of traveler's diarrhea if occurred (# days) | 3 weeks
Presence of symptoms associated with TD (cramps, nausea, fever, blood in the stools, vomiting, bloating, flatulence, visceral pain) | 3 weeks
Need for rescue medication | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Pontello, Prof., Principal Investigator — University of Milan, Milan, Italy
Locations (1):
- University of Milan, Milan, Italy